CLINICAL TRIAL: NCT01393145
Title: Multicenter, Phase III, Randomized, Open Label Study to Evaluate the Efficacy and Safety of a Fixed-dose Combination of Formoterol/Fluticasone and Salmeterol/Fluticasone in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Efficacy and Safety Study of Formoterol/Fluticasone and Salmeterol/Fluticasone in Patients With Moderate-to-severe COPD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-LLN-03(06/10)
Record Dates: First submitted 2011-03-09; First posted 2011-07-13 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: Chronic obstructive pulmonary disease (COPD); salmeterol; fluticasone; formoterol; FEV1; Moderate-to-severe
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate; Salmeterol Xinafoate; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: Combination Fluticasone /Formoterol 12/250 μg
- Group 2 (Active Comparator)
  Interventions: Drug: Seretide Diskus (salmeterol/fluticasone) 50/250 μg

INTERVENTIONS:
Drug: Combination Fluticasone /Formoterol 12/250 μg — Capsules containing Fumarate formoterol 12 µg + fluticasone propionate 250 µg dry powder for inhalation with aerocaps®
  Arms: Group 1
Drug: Seretide Diskus (salmeterol/fluticasone) 50/250 μg — Capsules containing salmeterol xinafoate 72.5 µg (equivalent to 50 µg of salmeterol) presented as powder for aspiration, packed in a plastic device in disk format, containing 60 doses
  Arms: Group 2

SUMMARY:
A study multicenter, phase III, randomized, open label study to evaluate the efficacy and safety of a fixed-dose combination of formoterol/fluticasone and salmeterol/fluticasone in patients with moderate-to-severe chronic obstructive pulmonary disease (COPD) that will enroll 336 subjects aged ≥ 40 years, smokers or former smokers, diagnosed with chronic obstructive pulmonary disease, classified as moderate chronic obstructive pulmonary disease or severe according to GOLD spirometric classification. The subjects will be allocated in 2 parallel groups and will receive the medicines of study, according of the randomization during a 24-week.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years;
2. Chronic obstructive pulmonary disease classified as moderate or severe according to GOLD guidelines (Global Initiative for Chronic Obstructive Lung Disease), with post-bronchodilator FEV1/FVC <0.70, and post-bronchodilator FEV1 <80% and ≥ 30% predicted;
3. Understanding and capacity to give written consent;
4. Smoker or ex-smoker of ≥ 10 pack-years [number of pack-years = number of daily cigarettes / 20 x number of years of smoking (eg t10 pack-years is equal to 20 cigarettes / day for 10 years, or 10 cigarettes per day within 20 years)].
5. Ability to fill out the patient's Diary
6. Ability to fill out the MRC dyspnea scale and questionnaires CAT and CDLM.

Exclusion Criteria:

1. Presence of clinically associate morbidities manifested according to the investigator that would interfere in the evaluation, for example: diabetes mellitus, congestive heart failure, coronary heart disease, chronic renal failure, liver failure, arrhythmia, hypothyroidism or hyperthyroidism;
2. Presence of neuro-psychiatric disorders of any kind;
3. Presence of mental retardation of any etiology;
4. Presence of pulmonary malformations, bronchiectasis, cystic fibrosis, bronchopulmonary hemosiderosis, ciliary dyskinesia, alveolitis, hypersensitivity, pulmonary vasculitis, sarcoidosis, tuberculosis or other lung diseases that might interfere with study assessments, as the investigator's discretion;
5. Subjects using immunosuppressive therapy, immunomodulatory agents, chemotherapy for allergy or any other immunotherapy;
6. Subjects using xanthine or acebrophylline;
7. Use within two months preceding the screening visit (V-2) of: anti-leukotrienes, immunoglobulins (including omalizumab), beta blockers, digitalis, itraconazole, amiodarone, antidepressants, monoamine oxidase inhibitors, tricyclic antidepressants, rifampin, oral contraceptives and coumarin ;
8. Current diagnosis of asthma;
9. Symptomatic coronary insufficiency;
10. Surgery for lung volume reduction and / or lung transplantation;
11. Need for long-term oxygen therapy (defined as the need for oxygen therapy ≥ 12 hours / day);
12. Pregnant or test β-HCG serum positive;
13. Lactating women;
14. Subject who uses more than 2 alcohol drinks a day or> 14 drinks a week;
15. Subject with a history of malignancy or ≤ 5 years> 5 years, but without documentation of remission / cure.
16. Illiterate or individuals who have limitation in understanding the use of devices as well as an inability to understand the questionnaires and diary that will be applied; Exception: subject illiterate, but capable of understanding regarding the use of the device, the questionnaires and diaries of the study and make available for relatives who can fill the diary study.
17. History of hypersensitivity to study drugs and rescue;
18. Any other disease or therapy that in the opinion of the investigator would jeopardize the subject or interfere with the objective of the study;
19. Subject with a history of ineffectiveness of formoterol fumarate, to fluticasone or salmeterol xinafoate;
20. Subject who participated in another study within 1 (one) year;
21. Pregnant women or those with positive serum β-HCG;
22. Radiological change is not compatible with COPD;
23. Clinically significant ECG changes, as reported by the investigator;
24. Any other disease, therapy or laboratory abnormality which in the opinion of the investigator would jeopardize the subject or interfere with the objective of the study;
25. Use of medications prescribed in the exclusion criteria for visit V -2.
26. Subjects who had an exacerbation during the standardization that required systemic corticosteroids and / or antibiotics or hospitalization will not be eligible for randomization.
27. Use of oral corticosteroids, anti-leukotrienes, immunoglobulins (including omalizumab), beta blockers, digitalis, amiodarone, itraconazole, antidepressants, monoamine oxidase inhibitors and tricyclic antidepressants during the period of standardization;
28. Any other disease or therapy that in the opinion of the investigator would jeopardize the subject or interfere with the objective of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Changes in pre-bronchodilator forced expiratory volume in first second (FEV1) | Comparative between baseline and week 24
  Changes of lung function parameter

SECONDARY OUTCOMES:
Changes in forced expiratory volume in first second, without bronchodilator | Week 0, 8, 16 and 24
  Changes of lung function parameter
Safety descriptive about occurence of adverse events, evaluation of results of clinical/physical examination and laboratory tests results | From baseline to week 24
  Collection of safety data throughout the whole study period
Changes in COPD Assessment Test (CAT) | Week 0, 8, 16 and 24
  Questionnaire